CLINICAL TRIAL: NCT00001118
Title: A Phase I/II Study of T-20, a Fusion Inhibitor, in HIV-1 Infected Children
Brief Title: Study of a New Anti-HIV Drug, T-20, in HIV-Infected Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: P1005; 11642 (Registry Identifier: DAIDS ES); ACTG P1005; PACTG P1005; T20-204
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Injections, Intravenous; Injections, Subcutaneous; Drug Therapy, Combination; HIV Protease Inhibitors; Membrane Fusion; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load; peptide T20
MeSH Terms: conditions — HIV Infections | interventions — Enfuvirtide

INTERVENTIONS:
Drug: Enfuvirtide

SUMMARY:
The purpose of this study is to determine the best dose of T-20, a new anti-HIV drug, to treat HIV-infected children.

T-20, unlike other anti-HIV medications, lessens the ability of HIV to infect certain cells (T cells) in the body. Doctors hope to better treat HIV by adding T-20 to anti-HIV drug combinations that include 1 or 2 nucleoside reverse transcriptase inhibitors (NRTIs) plus a nonnucleoside reverse transcriptase inhibitor (NNRTI) and/or a protease inhibitor (PI).

DETAILED DESCRIPTION:
T-20 is the first drug to be developed which specifically inhibits the function of the gp41 transmembrane glycoprotein. By inhibiting the essential protein-protein surface interaction, T-20 is able to block the process of virus-to-host cell membrane fusion. Combination antiretroviral regimens (reverse transcriptase inhibitors plus PIs) have benefited many HIV patients, but heavily pretreated patients often develop multi-drug resistance via multiple gene mutations. A pharmacologic agent, such as T-20, that is effective at an alternative point in the virus replication cycle will make a valuable addition to the treatment of HIV infection.

This Phase I/II open-label, dose-escalating, randomized study is divided into 2 parts. Patients may participate in Part A and/or Part B. Part A (single dosing): 12 patients are sequentially assigned to receive 1 of 3 doses of T-20 given once on Day 0 by SC injection into the abdomen, deltoid area, or anterior aspect of the thigh and once on Day 1 by IV infusion. Provided safety criteria are met, patients who complete Part A, or new enrollees who did not participate in Part A, enroll in Part B. Doses for Part B are determined by pharmacokinetic data obtained in Part A. [AS PER AMENDMENT 4/20/00: Current data has now projected a pediatric dose. Each child will move to chronic dosing in Part B provided the child has no Grade 3 or higher toxicity to study drug through Day 7 in Part A.] Part B (multiple dosing): Patients are randomly assigned to 1 of 3 dose cohorts to receive 24 weeks [AS PER AMENDMENT 12/7/00: 48 weeks] of treatment (optional extension to 48 weeks [AS PER AMENDMENT 12/7/00: 96 weeks]) with bid SC injections of T-20. Cohort 1 receives the dose identified in Part A (Dose 1) as the lowest dose that is well tolerated and that achieves the target trough plasma concentration. Cohort 2 receives the next higher dose from Dose 1 (Dose 2). Cohort 3 receives either Dose 1 or Dose 2, depending on the tolerability and antiviral activity of each dose. [AS PER AMENDMENT 4/20/00: Cohort 1 receives 30 mg/m2 SC bid (Dose 1); Cohort 2 receives 60 mg/m2 SC bid (Dose 2); and Cohort 3 receives Dose 1 or 2 SC bid.] On Day 7 of T-20 dosing, children begin a new antiretroviral therapy regimen chosen by the site investigator based on study parameters. (Abacavir and amprenavir are not allowed for this regimen.) [AS PER AMENDMENT 1/6/00: Abacavir and amprenavir are now allowed.] The first injection will be given in the clinic and a parent/guardian will be trained to give successive injections. [AS PER AMENDMENT 4/20/00: The 2 doses given prior to obtaining trough levels on Days 1 and 7 must be directly observed by medical personnel.] Patients undergo clinical and laboratory evaluations to monitor viral load, HIV-related symptoms, and pharmacokinetics at time points throughout the study. Patients participating in Part A are evaluated at the clinic on Days 0, 1, and 7. Patients participating in Part B are evaluated at the clinic 6 times during the first 3 weeks and then every 4 weeks through Week 24. [AS PER AMENDMENT 12/7/00: Patients participating in Part B are evaluated at the clinic 6 times during the first 3 weeks, every 4 weeks through Week 24, and then every 8 weeks through Week 48.]

ELIGIBILITY:
Inclusion Criteria

Children may be eligible for this study if they:

* Are 3 to 12 years old (consent of parent or guardian required).
* Are HIV-positive.
* Are receiving combination anti-HIV therapy. He/she must have been taking this combination for at least 16 weeks, and it must include either 2 NRTIs alone or 2 NRTIs plus either an NNRTI or a PI. (This study has been changed. This no longer has to be a child's first anti-HIV drug combination.)
* Have a viral load greater than 10,000 copies/ml while taking this anti-HIV drug combination.
* Have never received treatment with a PI or an NNRTI. (One or two doses are allowed.)
* Have never taken at least 1 NRTI.

Exclusion Criteria

Children will not be eligible for this study if they:

* Are receiving treatment for an opportunistic (AIDS-related) or serious bacterial infection at the time of study entry.
* Are receiving chemotherapy for cancer.
* Have certain serious diseases (other than HIV) or conditions.
* Have received or are currently receiving certain medications.
* Are pregnant.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24
Dates: Study Completion 2002-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Church, Study Chair; Coleen Cunningham, Study Chair
Locations (25):
- United States (24):
  - UCSD Med Ctr / Pediatrics / Clinical Sciences, La Jolla, California
  - Long Beach Memorial (Pediatric), Long Beach, California
  - Children's Hosp of Los Angeles/UCLA Med Ctr, Los Angeles, California
  - UCSF / Moffitt Hosp - Pediatric, San Francisco, California
  - Children's Hosp of Washington DC, Washington D.C., District of Columbia
  - Howard Univ Hosp, Washington D.C., District of Columbia
  - Univ of Florida Health Science Ctr / Pediatrics, Jacksonville, Florida
  - Univ of Miami (Pediatric), Miami, Florida
  - Tulane Univ / Charity Hosp of New Orleans, New Orleans, Louisiana
  - Children's Hosp of Boston, Boston, Massachusetts
  - Boston City Hosp / Pediatrics, Boston, Massachusetts
  - Baystate Med Ctr of Springfield, Springfield, Massachusetts
  - Univ of Massachusetts Med School, Worcester, Massachusetts
  - Children's Hosp of Michigan, Detroit, Michigan
  - Univ of Medicine & Dentistry of New Jersey / Univ Hosp, Newark, New Jersey
  - North Shore Univ Hosp, Great Neck, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Metropolitan Hosp Ctr, New York, New York
  - Harlem Hosp Ctr, New York, New York
  - SUNY Health Sciences Ctr at Syracuse / Pediatrics, Syracuse, New York
  - Bronx Lebanon Hosp Ctr, The Bronx, New York
  - Bronx Municipal Hosp Ctr/Jacobi Med Ctr, The Bronx, New York
  - Duke Univ Med Ctr, Durham, North Carolina
  - Med Univ of South Carolina, Charleston, South Carolina
- San Juan City Hosp, San Juan, Puerto Rico

REFERENCES:
- [Background] Kosel B, Church J, Cunningham C, Sista P, Aweeka F. Pharmacokinetics (PK) of selected doses of T-20, a fusion inhibitor, in HIV-1-infected children. 8th Conf Retro and Opportun Infect. 2001 Feb 4-8 (abstract no 726)
- [Result] Church JA, Cunningham C, Hughes M, Palumbo P, Mofenson LM, Delora P, Smith E, Wiznia A, Purdue L, Hawkins E, Sista P; PACTG P1005 Study Team. Pediatric AIDS Clinical Trials Group. Safety and antiretroviral activity of chronic subcutaneous administration of T-20 in human immunodeficiency virus 1-infected children. Pediatr Infect Dis J. 2002 Jul;21(7):653-9. doi: 10.1097/00006454-200207000-00010. PMID 12237598
- [Result] Soy D, Aweeka FT, Church JA, Cunningham CK, Palumbo P, Kosel BW, Sheiner LB; Pediatric AIDS Clinical Trial Group (PACTG) Study P1005 Investigators. Population pharmacokinetics of enfuvirtide in pediatric patients with human immunodeficiency virus: searching for exposure-response relationships. Clin Pharmacol Ther. 2003 Dec;74(6):569-80. doi: 10.1016/j.clpt.2003.09.002. PMID 14663459
- [Result] Church JA, Hughes M, Chen J, Palumbo P, Mofenson LM, Delora P, Smith E, Wiznia A, Hawkins E, Sista P, Cunningham CK; Pediatric AIDS Clinical Trials Group P1005 Study Team. Long term tolerability and safety of enfuvirtide for human immunodeficiency virus 1-infected children. Pediatr Infect Dis J. 2004 Aug;23(8):713-8. doi: 10.1097/01.inf.0000133045.45316.6a. PMID 15295220